CLINICAL TRIAL: NCT05208307
Title: Maintenance Therapy With Belantamab, Pomalidomide and Dexamethasone (BPd) in High-Risk Myeloma Patients: A Phase 2 Study With a Safety Run-In
Brief Title: Belantamab Mafodotin, Pomalidomide and Dexamethasone for the Treatment of High-Risk Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: GlaxoSmithKline (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003092; NCI-2021-08385 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship5382-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (belantamab mafodotin, pomalidomide, dexamethasone) (Experimental): Patients receive belantamab mafodotin IV over 30 minutes on day 1 of every other cycle, pomalidomide PO QD on days 1-21, and dexamethasone PO QD on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Belantamab Mafodotin; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Biological: Belantamab Mafodotin — Given IV
  Other Names: Belantamab Mafodotin-blmf; Blenrep; GSK2857916; J6M0-mcMMAF
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies the effect of belantamab mafodotin, pomalidomide, and dexamethasone in treating patents with high-risk myeloma. Belantamab mafodotin is a monoclonal antibody, called belantamab, linked to a chemotherapy drug, called mafodotin. Belantamab is a form of targeted therapy because it attaches to specific molecules on the surface of cancer cells, known as BCMA receptors, and delivers mafodotin to kill them. Chemotherapy drugs, such as pomalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Anti-inflammatory drugs, such as dexamethasone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving belantamab mafodotin, pomalidomide, and dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the combination of belantamab mafodotin, pomalidomide and dexamethasone (BPd) by assessing the >= complete response (CR) rates with BPd maintenance in patients with high-risk myeloma by International Myeloma Working Group (IMWG) criteria.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of BPd in patients with high-risk myeloma.

II. To determine the antitumor activity of BPd maintenance among high-risk myeloma patients.

TERTIARY/EXPLORATORY OBJECTIVE:

I. To evaluate the changes in microenvironment among patients receiving BPd maintenance.

OUTLINE:

Patients receive belantamab mafodotin intravenously (IV) over 30 minutes on day 1 of every other cycle, pomalidomide orally (PO) once daily (QD) on days 1-21, and dexamethasone PO QD on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Transplant-eligible myeloma patient that has undergone autologous stem cell transplant (ASCT) within one year of their diagnosis and has achieved >= partial response (PR) based on IMWG standard criteria. Patients will be enrolled within day 60-100 after ASCT
* Patient's with high-risk disease defined as

  * Presence of del(17p); t(4;14); t(14;16); t(14;20) by fluorescence in situ hybridization (FISH) or by cytogenetics (CTG)
  * Plasma cell leukemia at diagnosis with >= 20% circulating plasma cells on peripheral blood
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Participant must be >= 18 years of age
* Absolute neutrophil count (ANC) >=1.5 x 10^9/L (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Hemoglobin >= 8.0 g/dL (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Platelets >= 75 x 10^9/L (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (Isolated bilirubin >= 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Estimated glomerular filtration rate (eGFR) >= 30 mL/min/ 1.73 m^2 (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Spot urine (albumin/creatinine ratios) < 500 mg/g (56 mg/mmol) (performed within 28 days of initiation of protocol therapy unless otherwise specified)
* Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) OR
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

WOCBP refers to sexually mature female, regardless of sexual orientation or whether they have undergone tubal ligation, who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally menopausal for at least 24 consecutive months. A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

Nonchildbearing potential is defined as follows (by other than medical reasons):

* >= 45 years of age and has not had menses for > 1 year
* Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure

  * Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:
* Refrain from donating sperm PLUS either:
* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception/barrier as detailed below:

  * Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of < 1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females)

    * All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events [NCI-CTCAE], version 4.03) must be =< grade 1 at the time of enrolment except for alopecia
    * Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

* Participant must not have current corneal epithelial disease except mild changes in corneal epithelium
* Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis

  * Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
* Participant must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from multiple myeloma (MM) are eligible, provided they fulfil inclusion criteria
* Participant must not use contact lenses while participating in this study
* Participant must not be simultaneously enrolled in any interventional clinical trial
* Participant must not have used an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug
* Participant must not have had plasmapheresis within 7 days prior to first dose of study treatment
* Participant must not have received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs
* Participant must not have had major surgery =< 4 weeks prior to initiating study treatment
* Participant must not have any evidence of active mucosal or internal bleeding
* Participant must not have evidence of cardiovascular risk including any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of Screening
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system (NYHA, 1994)
  * Uncontrolled hypertension
* Participant must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment
* Participant must not have an active infection requiring treatment
* Known human immunodeficiency virus (HIV) infection, unless the participant can meet all of the following criteria:

  * Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load < 400 copies/mL
  * CD4+ T-cell (CD4+) counts >= 350 cells/uL
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the last 12 months
  * Note: consideration must be given to antiretroviral therapy (ART) and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment unless the participant can meet the following criteria:

  * RNA test negative
  * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative hepatitis C virus (HCV) RNA test after a washout period of at least 4 weeks
* Patients will hepatitis B will be excluded unless the following criteria can be met

  * SEROLOGY: Hepatitis B core antibody positive (HbcAb+), hepatitis B surface antigen negative (HbsAg-); SCREENING: Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) undetectable; DURING STUDY TREATMENT: Monitoring per protocol, antiviral treatment instituted if HBV DNA becomes detectable
  * SEROLOGY: HBsAg+ at screen or within 3 months prior to first dose; SCREENING: HBV DNA undetectable, highly effective antiviral treatment started at least 4 weeks prior to first dose of study treatment, baseline imaging per protocol, participants with cirrhosis are excluded; DURING STUDY TREATMENT: Antiviral treatment maintained throughout study treatment, monitoring and management per protocol

    * Note: presence of hep B surface antibody (HBsAb) indicating previous vaccination will not exclude a participant
* Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction
* Participant must not have any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures
* Diagnosed with smoldering MM, monoclonal gammopathy of undetermined significance, Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, amyloidosis or standard risk myeloma or secondary plasma cell leukemia
* High risk patients that did not achieve >= PR after stem cell transplant
* Participant has >= grade 2 peripheral neuropathy on clinical examination within 28 days before initiation of protocol therapy
* Participants must not be pregnant or lactating
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study
* Prior malignancy (within the last 5 years) except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Known hypersensitivity to acyclovir or similar anti-viral drug
* Known intolerance to steroid therapy
* Contraindication or prior intolerance to thromboembolic prophylaxis with aspirin, warfarin or low-molecular weight heparin
* Participants with known central nervous system (CNS) disease
* Poor tolerability or known allergy to any of the study drugs or compounds of similar chemical or biologic composition to dexamethasone, boron or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Up to 3 years
  Assessed per International Myeloma Working Group criteria (best response during maintenance therapy).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Toxicities of all patients will be tabulated as frequency and percentage. To evaluate the safety of the belantamab mafodotin, pomalidomide and dexamethasone (BPd) combination in the maintenance setting, proportion of safe patients will be estimated and its 95% confidence interval (CI) will be constructed by assuming binomial distribution. Adverse events will be graded using Common Terminology Criteria for Adverse Events (version 5.0).
Very good partial response rate with BPd maintenance | Up to 3 years
  Will be calculated as the proportion with 95% CI, assuming binomial distribution.
Stringent complete response rate with BPd maintenance | Up to 3 years
  Will be calculated as the proportion with 95% CI, assuming binomial distribution.
Overall response with BPd maintenance | Up to 3 years
  Will be calculated as the proportion with 95% CI, assuming binomial distribution.
Progression free survival | Up to 3 years
  Will be estimated with standard Kaplan-Meier method.
Duration of response | Up to 3 years
  Will be summarized with median and range.
Overall survival (OS) | Up to 3 years
  Will be estimated with standard Kaplan-Meier method. Both point and 95% CI of the median and other statistics (e.g., 6-month rate, 12-month rate, etc.) of OS will be calculated.
Minimal residual disease (MRD) negativity rate | Up to 3 years
  MRD detection will summarized using descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K. Nooka, MD,MPH,FACP, Principal Investigator — Emory University/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No